CLINICAL TRIAL: NCT03969537
Title: Telemedicine Follow-up for Patients With Cervical Dystonia Treated With Neurotoxin Injections
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The Allergan Foundation (Other)
Responsible Party: Principal Investigator, David Charles, Professor of Neurology, Vanderbilt University Medical Center
Other Study IDs: 190232
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Cervical Dystonia; Telemedicine
Keywords: Cervical Dystonia; Telemedicine; Telehealth
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Telemedicine: The patients selected to participate in the study are cervical dystonia (CD) patients who receive treatment at Vanderbilt University Medical Center, where the study takes place.
  Interventions: Other: Telemedicine follow-up visit

INTERVENTIONS:
Other: Telemedicine follow-up visit — Study participants will experience two telemedicine (live audio/video) visits.

SUMMARY:
Many cervical dystonia (CD) patients are limited in their ability to travel to the clinic for follow-up in between injection visits.

A telemedicine visit at the time of peak effectiveness of neurotoxin treatment may be valuable in informing the neurologist's choice of muscle selection and/or dose for the next injection visit. The primary objective of this study is to investigate both patient and physician satisfaction with the use of our telemedicine tool for this type of follow-up. After assessment of the subject, the neurologist will decide whether or not the telemedicine visit was informative to the upcoming injection visit. Subjects will answer questions at the end of the visit regarding their satisfaction with the follow-up and overall telemedicine communication. The principle investigator will complete a similar survey with additional questions about information gathered from the visit to assess the primary objective.

A secure video communications platform will be used for the visit, which will occur 2-4 weeks after the patient's last neurotoxin injection (around the time of peak effectiveness). The investigating neurologist will remotely assess the patient and make notes for the next injection visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any race, aged 18 and above
* Diagnosed with cervical dystonia and being treated with neurotoxin injections at Vanderbilt University Medical Center
* The subject, or if appropriate their medical decision maker, is willing and able to provide written informed consent.
* Email and internet access
* Personal computing device with audio/video capability

Exclusion Criteria:

* Subjects for whom participation in the study may cause medical harm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected to participate in the study are cervical dystonia (CD) patients who receive treatment at Vanderbilt University Medical Center, where the study takes place.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction with Telehealth | 4 months
  This questionnaire measures patient satisfaction with the telehealth visit scored 7 to 27

CONTACTS AND LOCATIONS:
Overall Officials: David Charles, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No